CLINICAL TRIAL: NCT04909515
Title: Naxitamab and Granulocyte-Macrophage Colony Stimulating Factor (GMCSF) and Isotretinoin for Consolidation of Patients With High-Risk Neuroblastoma in First Remission. An International, Open-Label,Uncontrolled, Single-Arm, Multicenter, Phase 2 Trial
Brief Title: Naxitamab and Granulocyte-Macrophage Colony Stimulating Factor (GMCSF) and Isotretinoin for Consolidation of Patients With High-Risk Neuroblastoma in First Remission.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to business priorities
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Neuroblastoma
Keywords: antibody; neuroblastoma; pediatric; naxitamab; first remission
MeSH Terms: conditions — Neuroblastoma | interventions — naxitamab; Granulocyte-Macrophage Colony-Stimulating Factor; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- naxitamab + GM-CSF + isotretinoin (Experimental): 8 cycles. Cycles 1+2 naxitamab + GM-CSF, cycles 3-5 naxitamab + GM-CSF + isotretinoin, cycles 6-8 isotretinoin
  Interventions: Drug: Naxitamab; Drug: GM-CSF; Drug: Isotretinoin

INTERVENTIONS:
Drug: Naxitamab — 3.0 mg/kg/day = 9.0 mg/kg/cycle
Drug: GM-CSF — 250 - 500 microgram/m2/day
Drug: Isotretinoin — 160 mg/m2/day

SUMMARY:
This is a single-arm, uncontrolled, international, multi-center, clinical,phase 2 trial, in patients ≥ 12 months of age with high-risk neuroblastoma in first remission. 120 patients will be enrolled to receive naxitamab + GM-CSF in combination with isotretinoin.

ELIGIBILITY:
Inclusion Criteria:

1. Documentet neuroblastoma at time of diagnosis defined as

   1. Histopathology of solid tumor biopsy, or
   2. Bone marrow aspirate or biopsy indicative of neuroblastoma plus high blood or urine catecholamine metabolite levels
2. Documented high-risk disease at time of initial diagnosis defined as

   1. MYNC-amplified at stage L2, M or MS (according to International Neuroblastoma Risk Group (INRG)) of any age or
   2. MYCN-nonamplified with stage M (according to INRG) and diagnosed at ≥ 18 months of age or
3. Patient must have completed frontline therapy, and achieved one of the following:

   1. verified complete response according to INRC (bone marrow positive minimal residual disease is allowed as assessed by RTqPCR at site) after completion of induction and consolidation with or without autologous stem cell transplantation
   2. Verified partial response according to INRC for primary site and soft tissue, bone, and bone marrow metastases at pre-autologous stem cell transplantation evaluation (i.e., myeloablative chemotherapy + autologous stem cell transplantation required as part of frontline regimen). Furthermore, bone marrow response must be with ≤ 5% tumor (of total nucleated cellular content) seen on any specimen from a bilateral bone marrow aspirate/biopsy and bone response must be with ≤ 3 areas of abnormal uptake on 123I-MIBG scintigraphy
4. Age ≥ 12 months at trial enrollment

Exclusion Criteria:

1. Verified progressive disease during induction or consolidation therapy
2. Any systemic anti-cancer therapy, including chemotherapy, within 3 weeks prior to enrollment
3. Autologous stem cell transplantation within 6 weeks prior to enrollment or ongoing toxicity caused by the autologous stem cell transplantation at the discretion of the Investigator
4. Therapeutic 131I-MIBG within 6 weeks prior to enrollment
5. Prior anti-GD2 therapy
6. Performance status of < 50% as per the Lansky scale (patients less than 16 years of age) or Karnofsky scale (patients aged 16 years or older)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival (PFS) | 2 years
  2-year PFS defined as the proportion of patients alive and without progressive disease (PD) or relapse 2 years after enrollment

SECONDARY OUTCOMES:
Progression free survival | 128 weeks
  Progression free survival (defined as time from enrollment until progressive disease/relapse or death, whichever comes first)
1-year progression free survival | 1 year
  1-year progression free survival defined as the proportion of patients alive and without progressive disease or relapse 1 year after enrollment
1-year and 2-year overall survival | 2 years
  1-year and 2-year overall survival defined as the proportion of patients alive 1 year and 2 years after enrollment, respectively
2-year event-free survival | 2 years
  2-year event-free survival, defined as the proportion of patients alive and without progressive disease, relapse, secondary malignancy or until last contact if no event occurred, 2 years after enrollment
Proportion of positive to negative minimal residual disease (MRD) after 2 cycles | 6 weeks
  Proportion of patients changing from minimal residual disease positive in bone marrow at enrollment (defined as patients assessed as minimal residual disease positive by RTqPCR of bone marrow at enrollment) to minimal residual disease negative at completion of Cycle 2
Proportion of patients with MD positive convert to MRD negative | 6 weeks
  Proportion of patients with disease in bone marrow at enrollment (i.e., minimal disease according to INRC) and convert to minimal residual disease negative (assessed by RTqPCR) at completion of Cycle 2

CONTACTS AND LOCATIONS:
Locations (9):
- Hong Kong Children's Hospital, Kowloon, Hong Kong
- Russia (3):
  - National Medical Research Center Pediatric Hematology, Oncology and Immunology n.a Dmitry Rogachev, Moscow
  - Research Institute of Pediatric Oncology ad Hematology of N.N. Blokhin National Medical Research Center of Oncology, Moscow
  - Raisa Gorbacheva Memorial Institute of Children Hematology and Transplantation Bone marrow Transplant Clinic, Saint Petersburg
- Singapore (2):
  - ICON Cancer Centre Novena, Singapore
  - KK Women's and Children's Hospital, Singapore
- South Korea (3):
  - Asan Medical Center Childrens Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Soeul